CLINICAL TRIAL: NCT03046511
Title: Comparison Between Post - Surgical Intraperitoneal Antibiotics Administration Vs. Intravenous Pre- Surgical Administration for the Prevention of Peritonitis After Insertion of Peritoneal Dialysis Catheter in Peritoneal Dialysis Patients
Brief Title: Peritonitis Prevention After Insertion of Peritoneal Dialysis Catheter.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Victor Frajewicki, MD, Head, Department of Nephrology and Hypertension, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMC-16-0067-CTIL
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Peritoneal Dialysis-associated Peritonitis; Peritoneal Dialysis Catheter Infection; Peritoneal Dialysis Complication
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraperitoneal (Experimental): One single dose of intraperitoneal Cefazolin 1000 mg via the recently inserted peritoneal catheter
  Interventions: Drug: Cefazolin
- Intravenous (Active Comparator): One single dose of intravenous Cefazolin 1000 mg one hour before catheter insertion
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — A post- procedure administration of Cefazolin will be compared with a pre-operative intravenous dose

SUMMARY:
An intraperitoneal implanted catheter is always necessary to perform Peritoneal Dialysis. Catheter insertion has been associated with infectious complication such as Exit Site Infection (ESI), Tunnel Infection and Peritonitis. The last one may lead to loss of the technique because the need of catheter removal. Most of international guidelines recommends the use of prophylactic antibiotics. Different protocols has been used, mostly intravenous single injection before the procedure. For the last 25 years our unit gives a single intraperitoneal dose of Cefazolin immediately after the catheter insertion. The aim of this study is compare the effect of a pre- operative IV dose os Cefazolin with a post- procedure intraperitoneal single dose administration of the same drug.

ELIGIBILITY:
Inclusion Criteria:

Subjects suffering from Chronic Kidney Disease, candidates to a intra- peritoneal catheter insertion

Exclusion Criteria:

Pregnancy; Active antibiotic treatment before the procedure; Known allergy to Cefazolin

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Peritonitis | 14 days
  Peritonitis asscociated catheter defined by cloudy effluent, high leukocyte count with neutrofilia

SECONDARY OUTCOMES:
Exit site infection | 14 days
  Infection defined by purulent discharge or local redness
Tunnel infection | 14 days
  Inflammation in the subcutaneous tract of the peritoneal catheter

CONTACTS AND LOCATIONS:
Overall Officials: Victor Frajewicki, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No